CLINICAL TRIAL: NCT06081686
Title: Phase I/II Study to Evaluate the Safety and Tolerability, Radiation Dosimetry and Pharmacokinetics, and Efficacy of [177Lu] Lu-XT033 Injection in Patients With Metastatic Prostate Cancer
Brief Title: Study of [177Lu] Lu-XT033 Injection in Patients With Metastatic Prostate Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sinotau Pharmaceutical Group (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XT-XTR010-1-01
Record Dates: First submitted 2023-08-25; First posted 2023-10-13 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; [177Lu]Lu-XT033 Injection
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase I:[177Lu]Lu-XT033 Injection (Experimental): During dose verification phase,Patients received [177Lu]Lu-XT033 Injection 1.11Gbq（30mCi）/1.85Gbq（50mCi）intravenously every 8 weeks (+/- 1 week) for a maximum of 6 cycles.
  Interventions: Drug: Phase I:[177Lu]Lu-XT033 Injection
- Phase II:[177Lu]Lu-XT033 Injection (Experimental): During dose expansion phase,patients received [177Lu]Lu-XT033 Injection at R2PD based on phase I.
  Interventions: Drug: Phase II:[177Lu]Lu-XT033 Injection

INTERVENTIONS:
Drug: Phase I:[177Lu]Lu-XT033 Injection — Six subjects were enrolled in the 1.11 Gbq (30 mCi) group of [177Lu] Lu-XT033 Injection. The last subject in this group completed the 4-week observation period after the first dose, With the consent of the Safety Monitoring Committee (SRC), 6 subjects were enrolled in the 1.85 Gbq (50 mCi) group. Both groups used 8 ± 1 weeks as the dosing interval .
  Arms: Phase I:[177Lu]Lu-XT033 Injection
Drug: Phase II:[177Lu]Lu-XT033 Injection — Patients received [177Lu]Lu-XT033 Injection every 8 weeks (+/- 1 week) for a maximum of 6 cycles.
  Arms: Phase II:[177Lu]Lu-XT033 Injection

SUMMARY:
This was a multicenter, open-label, phase I/II study to evaluate the safety and tolerability, radiation dosimetry and pharmacokinetic characteristics, and efficacy of [177Lu] Lu-XT033 injection in patients with metastatic prostate cancer, including a phase I study and a phase II extension study.

DETAILED DESCRIPTION:
The study for each participant consisted of a Screening period, a Treatment period and a Follow-up period.

In phase I,Six subjects were enrolled in the 1.11 Gbq (30 mCi) group of [177Lu] Lu-XT033 Injection. The last subject in this group completed the 4-week observation period after the first dose, With the consent of the Safety Monitoring Committee (SRC), 6 subjects were enrolled in the 1.85 Gbq (50 mCi) group. Both groups used 8 ± 1 weeks as the dosing interval for a total of 4 doses.In phase II,Subjects who met the inclusion and exclusion criteria were treated with [177Lu] Lu-XT033 injection at the recommended phase II dose（RP2D）.After Cycle 4 treatment and prior to Cycle 5 treatment, the investigator assessed the following criteria to determine whether:

The patient showed evidence of response (i.e. radiological, PSA, clinical benefit)

The patient had signs of residual disease on CT with contrast/MRI or bone scan

The patient had shown good tolerance to the [177Lu] Lu-XT033 Injection

If the patient met all of the criteria above and agreed to continue with additional treatment of [177Lu] Lu-XT033, the Investigator could administer 2 additional cycles. A maximum of 6 cycles of [177Lu] Lu-XT033 as allowed.

All subjects continued to undergo safety, tolerability, and efficacy assessments until the study-specified visit occurred or the subject was lost to follow-up or death whichever came first.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have the ability to understand and sign an approved informed consent form (ICF).
2. Patients must be >= 18 and <＝80 years of age.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Patients must have a life expectancy >6 months.
5. Patients must have histological, pathological, and/or cytological confirmation of prostate cancer.
6. Patients must be 68Ga-PSMA-11 Positron Emission Tomography (PET)/Computed Tomography (CT) scan positive。
7. Patients must have a castrate level of serum/plasma testosterone (<50 ng/dL or <1.7 nmol/L).
8. Patients must have received at least one NAAD (such as enzalutamide and/or abiraterone)； Patients must have been previously treated with at least 1, but no more than 2 previous taxane regimens.
9. Patients must have progressive mCRPC.
10. Patients must have adequate organ function。
11. Subjects of childbearing potential voluntarily use an effective method of contraception, such as condoms, oral or injectable contraceptives, Intra-uterine device（IUD）,etc., during treatment and within 6 months of the last use of the trial drug.

Exclusion Criteria:

1. Previous treatment with any of the following within 6 months of enrollment: Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Radium-223, hemi-body irradiation. Previous PSMA-targeted radioligand therapy is not allowed.
2. Known other malignancies.
3. Any systemic anti-cancer therapy (e.g. chemotherapy, immunotherapy or biological therapy within 28 days prior to day of enrollment.
4. Known hypersensitivity to the components of the study therapy or its analogs.
5. A superscan as seen in the baseline bone scan.
6. Patients with a history of Central Nervous System (CNS) metastases.
7. Uncontrolled, intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, cardiac arrhythmia, or other severe complications.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
For phase I:Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability])of [177Lu]Lu-XT033 on dose 1.11Gbq and 1.85Gbq | Through study completion, assessed up to 2 years.
  To evaluate the safety and tolerability of [177Lu]Lu-XT033 Injection assessed from the number and incidence of patients with adverse events using CTCAE v5.0 and physical examination, electrocardiogram and laboratory abnormality, etc
For phase I：Whole body and organ uptake of [177Lu]Lu-XT033 Injection | From the first subject enrolled to one week after the last subject completed the first dosing,assessed up to approximately 12 months
  Quantitate the absorbed radiation doses (expressed as Gy/MBq) of administered [177Lu]Lu-XT033 to kidneys, liver, lungs, spleen, bone/red marrow and salivary glands.
For phase I：Maximum plasma concentration (Cmax) of Lutetium [Lu 177] Lu-XT033 in patients. | From the first subject enrolled to one week after the last subject completed the first dosing,assessed up to approximately 12 months
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Cmax will be listed and summarized using descriptive statistics.
For phase I：Time of observed drug concentration occurrence (Tmax) of Lutetium [Lu 177] Lu-XT033 in patients. | From the first subject enrolled to one week after the last subject completed the first dosing,assessed up to approximately 12 months
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Tmax will be listed and summarized using descriptive statistics.
For phase I：Area Under plasma concentration-time Curve from time 0 to 168 hours (AUC0-168) of Lutetium [Lu 177] Lu-XT033 in patients. | From the first subject enrolled to one week after the last subject completed the first dosing,assessed up to approximately 12 months
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUC0-168 will be listed and summarized using descriptive statistics.
For phase II:Prostate-specific Antigen 50 (PSA50) Response | Through study completion, assessed up to 2 years.
  PSA50 response was defined as the proportion of participants who had a >= 50% decrease in PSA from baseline confirmed by a PSA measurement >= 4 weeks later.

SECONDARY OUTCOMES:
For phase I:Prostate-specific Antigen 50 (PSA50) Response | Through study completion, assessed up to 2 years.
  PSA50 response was defined as the proportion of participants who had a >= 50% decrease in PSA from baseline confirmed by a PSA measurement >= 4 weeks later.
For phase I/II:Best Percentage Change From Baseline in Prostate-specific Antigen (PSA) Level(PCWG3) | Through study completion, assessed up to 2 years.
  Best percentage change from baseline in PSA level was defined as the maximum percent decrease at any time post-baseline.
For phase I/II:Time to PSA progression | Through study completion, assessed up to 2 years.
  PSA progression was defined as: 1) Where a decline from baseline was documented, date that a >= 25% increase in PSA and an absolute increase of 2 ng/mL or more from the nadir was documented and confirmed by a second consecutive value obtained at least 3 weeks later. Rises in PSA within the first 12 weeks of the date of first dose were ignored; 2) Where no decline from baseline was documented, PSA progression was defined as a >= 25% increase from the baseline value along with an increase in absolute value of 2 ng/mL or more after 12 weeks from the date of first dose (without confirmation) as specified in the Prostate Cancer Clinical Trials Working Group 3 (PCWG3) guidelines.
For phase I/II:Radiographic Progression-free Survival (rPFS) | Through study completion, assessed up to 2 years.
  Radiographic progression-free survival (rPFS) was defined as the time (in months) from the date of enrollment to the date of radiographic disease progression per the Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria or death due to any cause.
For phase I/II:Overall Response Rate (ORR) | Through study completion, assessed up to 2 years.
  Overall Response Rate (ORR) was defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR). ORR was based on RECIST 1.1 response for patients with measurable disease at baseline.
For phase I/II: Duration of Response (DOR) | Through study completion, assessed up to 2 years.
  Duration of Response (DOR) was defined as the duration between the date of first documented Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) and the date of first documented radiographic progression or death due to any cause .
For phase I/II:Disease Control Rate (DCR) | Through study completion, assessed up to 2 years.
  Disease control rate (DCR) was defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) or Stable Disease (SD) according to RECIST v1.1.
For phase I/II:Health related quality of life(HRQOL) | Through study completion, assessed up to 2 years.
  Patient evaluation with questionnaires regarding Quality of Life .
For phase I/II:Time to First Symptomatic Skeletal Event (SSE) | Through study completion, assessed up to 2 years.
  Time to first Symptomatic Skeletal Event (SSE) was defined as the time (in months) from the date of enrollment to the date of the SSE or death from any cause. The SSE date was the date of first new symptomatic pathological bone fracture, spinal cord compression, tumor-related orthopedic surgical intervention, requirement for radiation therapy to relieve bone pain, or death due to any cause.
For phase I/II:Overall Survival (OS) | Through study completion, assessed up to 2 years.
  Overall Survival (OS) was defined as the time (in months) from the date of enrollment to the date of death due to any cause. If the patient was not known to have died, then OS was censored. The censoring date was date of the last study visit, or contact, until the cut-off date.
For phase II:Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability])of [177Lu]Lu-XT033 | Through study completion, assessed up to 2 years.
  To evaluate the safety and tolerability of [177Lu]Lu-XT033 Injection assessed from the number and incidence of patients with adverse events using CTCAE v5.0 and physical examination, electrocardiogram and laboratory abnormality, etc

CONTACTS AND LOCATIONS:
Overall Officials: Dingwei Ye, Principal Investigator — Fudan University; Zhi Yang, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (2):
- China (2):
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No